CLINICAL TRIAL: NCT06370832
Title: Inspiratory Muscle Training in Lung Transplant Candidates and Implications on Early Post-Transplant Outcomes: A Pilot and Feasibility Multicenter Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training in Lung Transplant Candidates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian National Transplant Research Program (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Ozmosis Research Inc. (Industry); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Vancouver General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-5171
Record Dates: First submitted 2024-03-04; First posted 2024-04-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Inspiratory Muscle Training
Keywords: Lung transplant candidates; Exercise training; Prehabilitation; Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Pre-lung transplant candidates will be randomized to one of two groups: (1) IMT + exercise training; or (2) exercise training alone.
Who Masked: Outcomes Assessor
Masking Description: Ascertainment of post-transplant clinical outcomes (including histopathology assessments) will be blinded by assessors to study group up to 3 months post-transplant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMT and exercise training group (Experimental): Participants in the IMT and exercise training group will perform twice daily 30-breath IMT sessions and exercise training sessions three times per week as part of their usual care during the pre-lung transplant phase. The exercise training is comprised of aerobic, resistance and flexibility training.
  Interventions: Other: IMT and exercise training group
- Usual care group (No Intervention): Participants in the usual care group will take part in the standard of care rehabilitation program provided during the waitlist phase prior to the transplant. Exercise training is performed at least three times per week for the duration of the waitlist period. The exercise training includes a combination of supervised in-person visits and home-based training that incorporates aerobic, resistance and flexibility training.

INTERVENTIONS:
Other: IMT and exercise training group — Participants will perform supervised exercise training per usual care and will be provided with a personalized prescription for an IMT program during the pre-transplant phase. Participants will perform two daily IMT sessions of 30 breaths (< 5 minutes/session) 5 days per week in their home environment or in-person visits. IMT intensity will be progressed weekly by 5-10% of the baseline maximal inspiratory pressure if the Borg Dyspnea score is < 7.
  Arms: IMT and exercise training group

SUMMARY:
Recovery after lung transplantation (LTx) may be complicated by prolonged mechanical ventilation (MV) and protracted intensive care unit (ICU) stay leading to immobilization and impaired health-related quality of life (HRQoL). In the critical care setting, diaphragm atrophy and weakness have been associated with difficulty weaning from MV, increased risk for readmission to hospital or ICU, and increased mortality. Increasing respiratory muscle strength by inspiratory muscle training (IMT) as part of pre-rehabilitation mitigates respiratory muscle dysfunction peri-operatively and may reduce the risk of post-operative complications. However, IMT is not widely used prior to LTx and the benefits of pre-operative IMT on post-transplant outcomes in LTx candidates have not been studied. Objectives: (1) To evaluate the feasibility of a multicenter randomized clinical trial of IMT in LTx candidates in terms of recruitment rate, retention, program adherence, and outcome ascertainment; (2) To establish the change in pre-transplant dyspnea perception, diaphragm structure and function, health related quality of life (HRQoL) and post-transplant intensive care unit (ICU), hospital and post-transplant 3-month outcomes with IMT relative to usual care group; and (3) To characterize the effect of pre-transplant IMT on peri-transplant diaphragm myofibrillar cross-sectional area (CSA), oxidative capacity, inflammatory markers and post-transplant diaphragm muscle thickness and function (UHN TGH site).

DETAILED DESCRIPTION:
Diaphragm atrophy at the time of initiating mechanical ventilation (MV) after solid organ transplantation and major surgery is associated with prolonged MV and higher hospital mortality. The incidence of diaphragm dysfunction after LTx is estimated to be up to 30%; post-transplant diaphragm dysfunction is associated with prolonged MV and hospitalization after LTx.

The American Thoracic Society/European Respiratory Society (2013) guidelines recommend further evaluation of inspiratory muscle training (IMT) combined with routine rehabilitation prior to major surgery. Pre-operative IMT in patients with even normal maximal inspiratory pressures (MIP) have been shown to decrease post-operative pulmonary complications and shorten hospitalization after cardio-thoracic surgery. However, pre-operative IMT is not commonly used for LTx candidates and its benefits are poorly researched. IMT may prove to be a simple pre-transplant intervention to prevent post-transplant morbidity and improve post-transplant functional status. The current focus is to investigate the impact of IMT on early post-lung transplant results while evaluating its effectiveness through a pilot multicenter randomized controlled trial.

Objectives: 1) To evaluate the feasibility of a multicenter randomized clinical trial of IMT in LTx candidates in terms of recruitment rate, retention, program adherence, and outcome ascertainment.

2) To establish the change in pre-transplant dyspnea perception, diaphragm structure and function, health related quality of life (HRQoL) and post-transplant intensive care unit (ICU), hospital and post-transplant 3-month outcomes with IMT relative to usual care group.

3) To characterize the effect of pre-transplant IMT on peri-transplant diaphragm myofibrillar cross-sectional area (CSA), oxidative capacity, inflammatory markers and post-transplant diaphragm muscle thickness and function (UHN TGH site).

Hypotheses: 1) It will be feasible to recruit LTx candidates into an IMT program RCT with a consent rate ≥ 30 %, enrolment rate of 2-3 patients per month at UHN and 1 patient per month at each other participating site, adequate outcome ascertainment (≥ 80%), and acceptable adherence (≥ 80% compliance with IMT sessions). 2) IMT will increase respiratory muscle endurance by 20% and improve exertional dyspnea and HRQoL in comparison to usual care over the pre-transplant period. IMT will be associated with greater hospital free days at 90 days. 3) pre-transplant IMT increases diaphragm myofibrillar CSA and post-LTx diaphragm thickness and maximal diaphragm thickening during inspiration in comparison to usual care. The improved mitochondrial respiration will occur concurrently with improvements in muscle fiber size, immune infiltration and oxidative stress.

The IMT and exercise training group (IMT group) will perform two daily IMT sessions of 30 breaths (< 5 minutes/session) during the pre-LTx period. IMT will start at 30% of MIP with a 5-10% weekly increase in training intensity guided by weekly MIP as tolerated (median weekly Borg dyspnea score < 7 during IMT until reaching 70% of MIP) and continued until LTx. In conjunction with their IMT program, IMT group participants will undergo exercise training at least three times per week as part of their usual care. The control group (exercise training group) will perform exercise training as part of their usual care three times per week for the duration of the waitlist period. The exercise regimen for both groups consists of aerobic, resistance, and flexibility training supervised by a physiotherapist approximately three times a week. The training includes a combination of in-person visits and home-based sessions. Both groups will also receive a respiratory endurance device to evaluate respiratory endurance throughout the trial.

IMT can improve respiratory muscle strength and endurance, potentially helping those who are candidates for LTx. In addition, studying patients undergoing LTx affords unique opportunities to investigate the mechanistic effects of IMT on diaphragm structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥ 18 years of age)
* Lung Transplant Candidates
* Participating in outpatient pulmonary rehabilitation (standard of care)
* Diagnosis of Interstitial Lung Disease or Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* Respiratory exacerbation within the last 1 month
* Neurologic or musculoskeletal conditions that may interfere with IMT or functional assessments (i.e. history of stroke, severe arthritis of hands)
* Insufficient English fluency to provide informed consent or to follow study protocols
* Any evidence of pneumothorax on recent imaging (< 6 months)
* Present ruptures of eardrums or infections leading to fluid behind ear drum
* Marked left or right ventricular end-diastolic volume and pressure overload on right heart catheterization or echocardiogram
* Severe osteoporosis with history of rib fractures
* Cardiac pacemaker or other electronic or magnetic body implant
* Individuals listed as rapidly deteriorating or inpatient at the time of eligibility assessment
* Individuals awaiting a re-transplant
* Inability of the patient to connect to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Study Recruitment According to Research Team Records | Over study recruitment period (approximately 2 years)
  Recruitment-success percentage in the study will be assessed based on research team study records.
Participant Retention in the Study According to Research Team Records | Over the study data collection period (from enrolment until 3 months post-transplant)
  Participant retention will be assessed by measuring participant follow-up throughout the study period, according to research team records. A retention rate of 80% or greater (in each group) has been established as the criteria to determine study feasibility.
Self-Reported Adherence to Inspiratory Muscle Training According to Participant IMT Diary | Over intervention period (from randomization until time of transplantation, up to maximum of 24 months)
  Adherence to inspiratory muscle training will be assessed via the IMT training diary completed by participants. Successful adherence will be defined as completion of ≥ 80% training sessions.
Adverse Events and IMT Training Side Effects Reported by Participants | Over intervention period (from randomization until time of transplantation, up to maximum of 24 months)
  Adverse events and training side-effects (e.g., muscle soreness) with inspiratory muscle training will be monitored through participant training diaries during the study intervention period. The research coordinator will review these diaries with participants on a weekly basis. Additionally, participants will be strongly encouraged to promptly inform the study team if they experience any challenges with IMT.
Inspiratory Muscle Training Satisfaction Questionnaire (IMT Group Only) | At 3 months post-transplant follow-up
  Participant satisfaction and motivation with the IMT intervention will be determined using a satisfaction questionnaire.

SECONDARY OUTCOMES:
Respiratory Muscle Endurance Test | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  Respiratory muscle endurance (measured in seconds) will be assessed at 30-50% of Maximum Inspiratory Pressure (MIP) using a manual threshold loading device (Powerbreathe Classic light resistance trainer)
Dyspnea Severity Assessed by Medical Research Council Dyspnea Scale | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  The Medical Research Council Dyspnea Scale will be used to assess the effect of breathlessness on daily activities. The scale comprises five statements that describe the range of respiratory dyspnea from none (Grade 1) to severe with difficulties performing self-care (Grade 5).
Qualitative Measures of Dyspnea Assessed by Qualitative Dyspnea Scale | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  The 18-point Qualitative Dyspnea Scale will be ascertained at each follow-up time point. Participants will be presented with a list of 18 qualitative descriptors of dyspnea experience and will be asked to rank their top three.
Mood Assessed by Depression, Anxiety, and Stress Scale | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  The Depression, Anxiety and Stress Scale (DASS-21) questionnaire has 21 items to assess mood (anxiety, depression, and stress). Each statement for the three domains is given a score of 0 (not applicable) to 3 (applicable most of the time) with scores categorized as follows: Normal, Mild, Moderate, Severe, and Extremely Severe.
Health-Related Quality of Life Assessed by St. George's Respiratory Questionnaire | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  Health-related Quality of Life (HRQL) will be assessed through the St. George's Respiratory Questionnaire (SGRQ) and consists of three domains (symptoms, activity and impacts) and total score. The SGRQ has a range of scores from 0 to 100 with higher scores signifying worse HRQL.
Respiratory Muscle Strength Assessed by Maximal Inspiratory Pressure | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), time of liberation from mechanical ventilation, and 3 months post-transplant
  Respiratory muscle strength will be quantified as Maximal Inspiratory Pressure (MIP), evaluated using a respiratory muscle trainer (PowerBreathe KH2).
Physical Activity and Exercise Behaviors Assessed by International Physical Activity Questionnaire | Change from baseline at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) will be used to measure physical activity levels in study participants. The questionnaire consists of seven questions to capture average daily time spent sitting, walking, and engaging in moderate and vigorous physical activity over the last seven days. The IPAQ-SF provides an overall physical activity level of participants based on their Metabolic Equivalent Task minutes per week.
Pulmonary Function Testing (Spirometry) | Baseline, 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  Clinical charts will be reviewed to obtain results from spirometry assessments including Forced Vital Capacity (FVC), and Forced Expiratory Volume in the first second (FEV1).
Aerobic Endurance Assessed by the Six-Minute Walk Test | Baseline, 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  Clinical rehabilitation charts will be reviewed to document aerobic endurance as assessed by distance walked during the Six-Minute Walk Test.
Physical Function Assessed by the Short Physical Performance Battery | Baseline, 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), and 3 months post-transplant
  Clinical rehabilitation charts will be reviewed to document physical function as assessed by the Short-Physical Performance Battery, which evaluates balance, gait speed, and ability to rise from a chair 5 times.
Pre-Transplant Hospitalizations | From baseline up until the time of admission for the index transplant hospitalization (up to 24 months total)
  Clinical charts will be reviewed to document any hospitalizations and ICU admissions before the time of transplantation.
Peri-Transplant Mechanical Ventilation Bridging | Peri-operative period, from time of index transplant hospital admission to time of transplant surgery (up to 24 months total)
  Clinical charts will be reviewed to determine whether mechanical ventilation or extracorporeal membrane oxygenation (ECMO) were required as a bridge to transplantation.
Post-Transplant Duration of Mechanical Ventilation (Days) | From time of transplant surgery to the time of liberation from mechanical ventilation (up to 3 months total)
  Clinical charts will be reviewed to determine the duration of mechanical ventilation required following transplantation surgery, measured in days.
WIND Weaning Classification | At the time of liberation from mechanical ventilation following transplant surgery (up to 3 months total).
  The WIND weaning classification (short, difficult, or prolonged) will be ascertained by ICU staff at the time of liberation from mechanical ventilation based on the number of spontaneous breathing trials and weaning difficulty.
Post-Transplant Hospital Length of Stay (Days) | From time of transplant surgery to the time of discharge from hospital (up to 3 months total).
  Clinical charts will be reviewed to determine the length of stay in hospital following transplant surgery, measured in days.
Post-Transplant Discharge Disposition | Time of discharge from index transplant hospitalization (up to 3 months total).
  Clinical charts will be reviewed to determine participants' discharge disposition from the index transplant hospitalization (e.g., home, inpatient rehabilitation, long-term care).
Primary Graft Dysfunction | Up to 72 hours post-transplant
  Clinical charts will be reviewed to determine the presence and severity of primary graft dysfunction following transplant surgery.
Post-Transplant Mortality | Up to 90 days (3 months) post-transplant
  Clinical charts will be reviewed to document post-transplant mortality and etiology.
Days Alive and at Home at 90 Days (DAAH90) | Up to 90 days (3 months) post-transplant
  Clinical charts will be reviewed to determine the number of days participants are alive and at home at 90 days post-transplant.

OTHER OUTCOMES:
Diaphragm Thickness and Thickening Fraction Assessed by Ultrasound | Change from baseline to all on-site visits at 4 weeks, 8 weeks, 12 weeks, every 3 months until lung transplant (up to 24 months total), time of liberation from MV, and 3 months post-transplant
  The right hemi-diaphragm thickness and thickening fraction will be measured using a 13 Megahertz ultrasound transducer. Bright-mode (B-mode) ultrasound will be used to visualize the diaphragm and motion-mode (M-mode) will be utilized to assess the amplitude of the cranio-caudal diaphragmatic excursion during quiet and deep breathing. Diaphragm thickness will be measured in M-mode with a 5-13 MHz linear transducer over the apposition zone, near the costophrenic angle, from the most superficial hyperechoic line (pleural line) to the deepest hyperechoic line (peritoneal line).
Histopathology Analyses of Diaphragm Biopsies (Optional) | At the time of lung transplantation, up to maximum of 24 months after randomization
  Participants will have the option of consenting to diaphragm biopsies collected during the transplant surgery. Biopsies (50 mg) will be procured from the anterolateral region of the right costal hemi-diaphragm midway between the origin and insertion. A portion of the tissue sample (20mg) will be fixed in formalin for histopathology analyses including assessing fibre type distribution, fibre type-specific cross-sectional area, immune infiltration, oxidative capacity, and fibrosis using light microscopy.
Biochemical Analyses of Diaphragm Biopsies (Optional) | At the time of lung transplantation, up to maximum of 24 months after randomization
  A second tissue portion (20mg) will be flash frozen in liquid nitrogen to assess mitochondrial content (via western blotting) and signaling cascades to examine atrophic signaling cascades using polymerase chain reactions.
Mitochondrial Respirometry Analyses of Diaphragm Biopsies (Optional) | At the time of lung transplantation, up to maximum of 24 months after randomization
  The final tissue portion (10 mg) will be used for live assessments of mitochondrial function using the Oroboros O2K High Resolution Respiratory system on the day of transplantation, as quickly after biopsy collection as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Rozenberg, MD, PhD, Principal Investigator — University Health Network/University of Toronto
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - University Health Network, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weill D, Benden C, Corris PA, Dark JH, Davis RD, Keshavjee S, Lederer DJ, Mulligan MJ, Patterson GA, Singer LG, Snell GI, Verleden GM, Zamora MR, Glanville AR. A consensus document for the selection of lung transplant candidates: 2014--an update from the Pulmonary Transplantation Council of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2015 Jan;34(1):1-15. doi: 10.1016/j.healun.2014.06.014. Epub 2014 Jun 26. PMID 25085497
- [Background] Hook JL, Lederer DJ. Selecting lung transplant candidates: where do current guidelines fall short? Expert Rev Respir Med. 2012 Feb;6(1):51-61. doi: 10.1586/ers.11.83. PMID 22283579
- [Background] Fuehner T, Kuehn C, Welte T, Gottlieb J. ICU Care Before and After Lung Transplantation. Chest. 2016 Aug;150(2):442-50. doi: 10.1016/j.chest.2016.02.656. Epub 2016 Mar 4. PMID 26953218
- [Background] Christie JD, Kotloff RM, Ahya VN, Tino G, Pochettino A, Gaughan C, DeMissie E, Kimmel SE. The effect of primary graft dysfunction on survival after lung transplantation. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1312-6. doi: 10.1164/rccm.200409-1243OC. Epub 2005 Mar 11. PMID 15764726
- [Background] Adler D, Dupuis-Lozeron E, Richard JC, Janssens JP, Brochard L. Does inspiratory muscle dysfunction predict readmission after intensive care unit discharge? Am J Respir Crit Care Med. 2014 Aug 1;190(3):347-50. doi: 10.1164/rccm.201404-0655LE. No abstract available. PMID 25084264
- [Background] Sklar MC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Rittayamai N, Harhay MO, Reid WD, Tomlinson G, Rozenberg D, McClelland W, Riegler S, Slutsky AS, Brochard L, Ferguson ND, Goligher EC. Association of Low Baseline Diaphragm Muscle Mass With Prolonged Mechanical Ventilation and Mortality Among Critically Ill Adults. JAMA Netw Open. 2020 Feb 5;3(2):e1921520. doi: 10.1001/jamanetworkopen.2019.21520. PMID 32074293